CLINICAL TRIAL: NCT02457312
Title: The Effect of 7 Days of Letrozole Pretreatment Combined With Misoprostol on the Placental and Decidual Tissues
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lee Chi Yan Vivian, Associate Consultant, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 12-077
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole group (Active Comparator): Letrozole 10 mg daily for 7 days before suction evacuation
  Interventions: Drug: Letrozole
- Placebo group (Placebo Comparator): Placebo tablets (look identical to letrozole tablets) daily for 7 days before suction evacuation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — letrozole 10 mg daily for 7 days before suction evacuation
  Other Names: Letrozole group
  Arms: Letrozole group
Drug: Placebo — placebo tablets which look identical to the letrozole tablets for 7 days before suction evacuation
  Other Names: Placebo group
  Arms: Placebo group

SUMMARY:
The present study aims at studying the effect of letrozole in early pregnancy in placenta and decidua including the progesterone receptor and the apoptotic factors.

DETAILED DESCRIPTION:
Twenty healthy subjects requesting legal surgical abortion up to 63 days gestation will be recruited for this study. They will be randomized to receive either placebo tablets or letrozole 10 mg daily for 7 days before suction evacuation. Suction evacuates which include the placenta and some decidua collected by the procedure in these 20 subjects will be used for the laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age should be up to 63 days. An ultrasound assessment would be performed to confirm the gestation.
* The woman is willing and able to participate after the study has been explained
* Age >18 years old

Exclusion Criteria:

* Criteria for prospective exclusion

Any indication of past or present ill health will be considered a contraindication for recruitment to the study. In particular, subjects should not be recruited if any of the following conditions is present:

1. multiple pregnancies
2. uterine fibroids
3. any significant medical disorder
4. intrauterine contraceptive device in situ
5. contra-indications to the use of letrozole or misoprostol

   * Criteria for exclusion from a secondary analysis

Situation in which subjects who have been formally admitted to the study could be excluded from a secondary analysis include:

1. the use of drugs other than those prescribed by the investigator for the treatment of possible therapy-related side-effects especially drugs with prostaglandin synthetase inhibitory activity such as salicylates, indomethacin or mefenamic acid
2. any violation of the study protocol
3. essential data missing from the subject's records making it impossible to judge the treatment outcome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The expression of progesterone receptors and apoptotic factors in the placental and decidual cells by immunostaining. | 8 days

SECONDARY OUTCOMES:
Apoptosis in the placental and decidual cells as demonstrated by TUNEL assay. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Vivian CY Lee, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China